CLINICAL TRIAL: NCT04646889
Title: A Phase 1, Pharmacokinetic and Pharmacodynamic Study of AR882 in Adult Volunteers With Various Degrees of Renal Impairment
Brief Title: Pharmacokinetic Study of AR882 in Subjects With Various Degrees of Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arthrosi Therapeutics (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AR882-104
Record Dates: First submitted 2020-11-18; First posted 2020-11-30 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Renal Impairment (Experimental): Subjects with various degrees of renal impairment
  Interventions: Drug: AR882 Single Dose; Drug: AR882 Multiple Dose
- Normal Renal Function (Experimental): Subjects with normal renal function
  Interventions: Drug: AR882 Single Dose; Drug: AR882 Multiple Dose

INTERVENTIONS:
Drug: AR882 Single Dose — A single dose of AR882
Drug: AR882 Multiple Dose — AR882 taken once daily for 14 days

SUMMARY:
This is a 2-segment, multi-center, phase 1, open-label, study evaluating the pharmacokinetics and pharmacodynamics of AR882 in subjects with various degrees of renal impairment.

ELIGIBILITY:
Inclusion Criteria:

All Subjects:

* Males and non-pregnant, non-lactating females
* Body weight no less than 50 kg
* sUA greater than or equal to 4.0 mg/dL

Renal Impaired Subjects:

• History of chronic renal impairment (> 6 months)

Exclusion Criteria:

All Subjects:

* Malignancy within 5 years, except for successfully treated basal or squamous cell carcinoma of the skin
* History of cardiac abnormalities
* Active peptic ulcer disease or active liver disease
* History of kidney stones

Renal Impaired Subjects:

• Requires dialysis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-01-14 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-06-27 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) for plasma following a single dose of AR882 in subjects with renal impairment and normal renal function | 6 days
Time to maximum plasma concentration (Tmax) following a single dose of AR882 in subjects with renal impairment and normal renal function | 6 days
Maximum plasma concentration (Cmax) following a single dose of AR882 in subjects with renal impairment and normal renal function | 6 days
Terminal half-life (t 1/2) following a single dose of AR882 in subjects with renal impairment and normal renal function | 6 days
Amount excreted (Ae) into urine following a single dose of AR882 in subjects with renal impairment and normal renal function | 6 days
Renal clearance (CLr) following a single dose of AR882 in subjects with renal impairment and normal renal function | 6 days
AUC for plasma following multiple doses of AR882 in subjects with renal impairment and normal renal function | 15 days
Tmax following multiple doses of AR882 in subjects with renal impairment and normal renal function | 15 days
Cmax following multiple doses of AR882 in subjects with renal impairment and normal renal function | 15 days
t 1/2 following multiple doses of AR882 in subjects with renal impairment and normal renal function | 15 days

SECONDARY OUTCOMES:
Incidence of Adverse Events, changes in laboratory, electrocardiogram, and vital signs following a single dose of AR882 in subjects with renal impairment and normal renal function | 14 days
Incidence of Adverse Events, changes in laboratory, electrocardiogram, and vital signs following multiple doses of AR882 in subjects with renal impairment and normal renal function | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Hingorani, MD, PhD, MBA, Study Director — Arthrosi Therapeutics
Locations (4):
- United States (2):
  - Arthrosi Investigative Site, Orlando, Florida
  - Arthrosi Investigative Site, Dallas, Texas
- New Zealand (2):
  - Arthrosi Investigative Site, Auckland
  - Arthrosi Investigative Site, Christchurch

IPD SHARING:
Plan to Share IPD: No